CLINICAL TRIAL: NCT03645161
Title: Comparison Between Local and Imported Skin Prick Testing Result of Rat and Mouse Allergen Extracts in Respiratory Allergy Patients
Brief Title: Comparison Between Local and Imported Skin Prick Testing Result of Rat and Mouse Allergen Extracts
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Nualanong Visitsunthorn, Professor, Mahidol University
Allocation: Non-Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: 789/2560 (EC 2)
Record Dates: First submitted 2018-08-22; First posted 2018-08-24 (Actual); Last update posted 2019-08-14 (Actual); Status verified 2019-08

CONDITIONS: Allergic Rhinitis Due to Animal Hair and Dander

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Local rat and mouse skin test (Active Comparator): All patients receive local skin prick test for mouse and rat. The result were recorded and compared to the imported one.
  Interventions: Diagnostic Test: rat and mouse skin test
- Imported rat and mouse skin test (Active Comparator): All patients receive imported skin prick test for mouse and rat. The result were recorded and compared to the local one.
  Interventions: Diagnostic Test: rat and mouse skin test

INTERVENTIONS:
Diagnostic Test: rat and mouse skin test — Comparison between local and imported skin prick testing result of rat and mouse allergen extracts in respiratory allergy patients

SUMMARY:
In respiratory allergy patients, skin prick test results of local rat and mouse allergen extracts are not significant different from imported ones

DETAILED DESCRIPTION:
Many researches proposed that rodent deteriorate symptoms in patients with respiratory allergy who sensitized. The test that can identify rodent sensitization will be very useful. The investigators found lots of problems from imported mouse and rat allergen extract, eg. expensive cost and hard to find importing agency in Thailand. Making own local allergen extract will be the good solution for the country. This study aim to compare the results of locally rat and mouse allergen to imported ones.

ELIGIBILITY:
Inclusion Criteria:

* Patients age 3 to 60 years old who diagnosed with asthma or allergic rhinitis
* Patient must not take these following medication at least 7 days before doing the skin prick test: antihistamine, oral corticosteroid (more than 20 mg/day of prednisolone), topical steroid that was apply on skin test area.

Exclusion Criteria:

* Pateints who have other chronic underlying disease e.g. obesity, heart disease and liver disease
* Patient with allergic asthma who is still uncontrollable.
* Patient with active severe atopic dermatitis
* Patient who are pregnant or in lactating period
* Patient or parent deny to join in the study

Ages: 3 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 230 (Actual)
Dates: Start 2018-05-30 (Actual); Primary Completion 2019-05-30 (Actual); Study Completion 2019-07-30 (Actual)

PRIMARY OUTCOMES:
Comparison between local and imported skin prick testing result of rat and mouse allergen extracts in respiratory allergy patients | 1 year
  Compare the results of locally rat and mouse allergen to imported ones.

CONTACTS AND LOCATIONS:
Overall Officials: Nualanong Visitsunthorn, MD, Principal Investigator — Department of Pediatrics, Siriraj hospital, Mahidol University
Locations (1):
- Siriraj Hospital. Mahidol University, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Undecided
publication